CLINICAL TRIAL: NCT06963931
Title: Change 4 Better (C4B): A Smartphone App to Address Problem Gambling
Brief Title: Change 4 Better (C4B)
Acronym: C4B
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Mohegan Sun Problem Gambling Treatment Fund (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000039709
Record Dates: First submitted 2025-05-01; First posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Problem Gambling
Keywords: Problem gambling; mobile app

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Change4Better (C4B) app plus Treatment As Usual (TAU) (Experimental): Participants will work with a mobile app that teaches skills for managing gambling. They will learn skills that may help with cognitive distortions related to gambling - for example, how seemingly unrelated events might be related to gambling outcomes. Participants will be taught how to use the mobile app by a staff member and will be asked to spend about 8 hours using the program (approximately 30-45 minutes per module) at home and will be encouraged to complete over the course of 12 weeks. Monthly follow-up will occur for an additional 12 weeks at which time the mobile app will also be available to participants.
  Interventions: Behavioral: Change4Better (C4B) mobile app
- Treatment As Usual (TAU) (No Intervention): Treatment As Usual (TAU) will consist of standard services provided at outpatient clinics within the Bettor Choice Programs. TAU will be tailored to the participants needs, and generally includes individual and/or group therapy sessions. Sessions will generally last for 1 hour one time per week for the first 12 weeks and include issues such as:
  * Teaching about the treatment program at the clinic
  * Teaching important ideas about recovery
  * Increasing knowledge about specific problems participants may have about with gambling
  * Demonstrating new ways of coping with skills designed to fit participants lifestyle.

INTERVENTIONS:
Behavioral: Change4Better (C4B) mobile app — The content of the C4B app is designed to teach key CBT strategies to address gambling behaviors. The content targets concerns that people with gambling problems often experience (gambling debts, cognitive distortions related to gambling - for example, how unrelated events might be related to gambling outcomes). We have designed the content such that people using the app can see the pattern of progress, identify mistakes and setbacks, and learn from common experiences of people with gambling disorder
  Arms: Change4Better (C4B) app plus Treatment As Usual (TAU)

SUMMARY:
The purpose of this research study is to determine the effectiveness of the Change4Better (C4B) mobile app at reducing the severity of problem gambling as compared to standard treatment as usual (TAU).

DETAILED DESCRIPTION:
This study is a 6-month randomized clinical trial for individuals with a gambling disorder enrolled in or seeking treatment for problem gambling at an outpatient treatment facilities affiliated with the Bettor Choice Gambling Treatment Programs in Connecticut. The purpose is to evaluate the feasibility and efficacy of a cognitive behavioral therapy-based mobile app (Change4Better; C4B), as an adjunct to treatment as usual (TAU) in community-based outpatient treatment programs. Eligible participants will be randomly assigned to receive either: (1) standard treatment as usual (TAU) or (2) TAU plus access to the Change4Better (C4B) mobile app. TAU will consist of standard services provided at outpatient clinics within the Bettor Choice Programs. Clinicians providing TAU within the Bettor Choice Program will not be participants in the research trial, and they will not be asked to perform any additional duties outside of their typical services. Participants assigned to C4B will receive TAU plus access to the C4B mobile app, which they can access as often as desired using their own device. The C4B mobile app will be managed by the Yale research team.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older;
2. able to speak, read and write in English;
3. report gambling in the past month (28 days);
4. meet DSM-5 criteria for gambling disorder within past 12 months as determined by the Structured Clinical Interview for Pathological Gambling - DSM-5 version (SCI-PG-DSM);
5. at least mild gambling severity as measured by GSAS (Total >8)
6. seeking or currently enrolled in treatment for gambling; if seeking treatment, must be deemed appropriate for outpatient level of care by treatment facility clinical team
7. own a smartphone with internet access.

Exclusion Criteria:

1. unwilling or unable to provide informed consent due to severe cognitive impairment or inability to read;
2. deemed to have current untreated psychosis or mania;
3. active suicidal ideation;
4. physical dependence on opioids and/or alcohol requiring medical detoxification.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in gambling symptom severity | Baseline to 6 months
  Change in gambling symptom severity as measured monthly by the Gambling Symptom Assessment Scale (G-SAS) from baseline to 6 months. Each item is scored on a 5-point scale from 0 (no symptoms) to 4 (extreme symptoms). The total score ranges from 0 to 48.

SECONDARY OUTCOMES:
App engagement-Days Used | Randomization through week 12
  Measured by number of days participants used the app
App engagement- Topics completed | Randomization through week 12
  Measured by number of topics completed by participants
App engagement- Practice exercises | Randomization through week 12
  Measured by number of practice exercises completed
App engagement- Weekly usage | Randomization through week 12
  Measured by average number of minutes per week participants used the app
App engagement- Total time | Randomization through week 12
  Measured by total time participants spent in the app

CONTACTS AND LOCATIONS:
Overall Officials: Brian Kiluk, PhD, Principal Investigator — Yale Universaity
Locations (4):
- United States (4):
  - CommuniCare, New Haven, Connecticut
  - Connecticut Renaissance, Norwalk, Connecticut
  - United Community & Family Services, Norwich, Connecticut
  - MCCA, Waterbury, Connecticut

IPD SHARING:
Plan to Share IPD: No